CLINICAL TRIAL: NCT04081610
Title: Phase I Clinical Trial to Evaluate the Safety and Tolerability of Lagricel® Ofteno Multi-dose Ophthalmic Solution Compared to Lagricel® Ofteno Single Dose on the Ocular Surface of Clinically Healthy Subjects
Brief Title: Clinical Trial to Evaluate the Safety and Tolerability of Lagricel® Ofteno Multi-dose Ophthalmic Solution
Acronym: PRO-037
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOPH037-0119/I
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-03

CONDITIONS: Dry Eye
Keywords: Dry eye; eye lubricant; sodium hyaluronate
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: single-center, controlled, parallel group, open, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lagricel® Ofteno Multidose (Experimental): Lagricel® Ofteno Multidose 0.4% hyaluronate. Ophthalmic solution. Laboratorios Sophia
  Interventions: Drug: lagricel ofteno multidose
- Lagricel® Ofteno Single dose (Active Comparator): Lagricel® Ofteno single dose. 0.4% hyaluronate. Ophthalmic solution. Laboratorios Sophia
  Interventions: Drug: lagricel ofteno single dose

INTERVENTIONS:
Drug: lagricel ofteno multidose — * Dosage: 1 drop 4 times a day per 7 days, both eyes
  * Route of administration: Ophthalmic
  Other Names: sodium hyaluronate 0.4%
  Arms: Lagricel® Ofteno Multidose
Drug: lagricel ofteno single dose — * Dosage: 1 drop 4 times a day per 7 days, both eyes
  * Route of administration: Ophthalmic
  Other Names: sodium hyaluronate 0.4%
  Arms: Lagricel® Ofteno Single dose

SUMMARY:
Study design: Phase I clinical trial, single-center, controlled, parallel group, open, randomized.

Number of subjects: n = 34 evaluable subjects, 17 evaluable subjects per group (both eyes).

Estimated duration of the study: 5 months

Therapeutic indication: Eye lubricant Use: Dry Eye

Objective:To evaluate the safety and tolerability of Lagricel® Ofteno multidose manufactured by Laboratorios Sophia on the ocular surface of clinically healthy subjects.

Hypothesis:

H0 = Lagricel® Ofteno multidose ophthalmic solution has a safety and tolerability profile similar to Lagricel® Ofteno single dose in healthy subjects.

H1 = Lagricel® Ofteno multidose ophthalmic solution has a different safety and tolerability profile than Lagricel® Ofteno single dose in healthy subjects.

Main inclusion criteria: Clinically healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* To be clinically healthy
* To have the ability to voluntarily grant your signed informed consent
* To have the willingness to comply with scheduled visits treatment plan and other study procedures
* Women in reproductive age should ensure the continuation (initiated ≥ 30 days prior to the signing of the informed consent) to use a hormonal contraceptive method or intrauterine device during the study period.
* To have a better corrected visual acuity of 20/30 or better in both eyes.
* To have vital signs in normal parameters.
* To have an intraocular pressure between ≥10 and ≤ 21 mmHg.

Exclusion Criteria:

* To be user of ophthalmic topical products of any kind.
* To be user of medicines, or herbal products, by any other route of administration.
* In the case of women: being pregnant, breastfeeding or planning to get pregnant in the study period.
* Having participated in clinical research studies 90 days prior to inclusion in this study.
* Having previously participated in this same study.
* To be a user of contact lenses and can not suspend their use during the study.
* Having initiated the use of hormonal contraceptives or intrauterine devices, 30 days prior to inclusion in the present study.
* To have a history of any chronic degenerative disease.
* Having inflammatory or infectious disease, active at the time of admission to the study.
* Having injuries or unresolved injuries at the time of admission to the study.
* Having a history of any type of eye surgery.
* Having undergone surgical procedures, not ophthalmological, in the last 3 months.
* To be or to have an immediate family member (for example: spouse, parent / legal guardian, brother or child) who is part of the research site staff or the sponsor who participates directly in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Biomedical research G & LS de RL de CV, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
Laboratorios Sophia, S.A. de C.V., serving as the sponsor of the study, assumes full responsibility for its function and retains exclusive ownership rights over the results of the study.
  The principal investigator undertakes not to publish or communicate data collected from the study, unless there is prior written agreement of Laboratorios Sophia, S.A. de C.V.

REFERENCES:
- [Derived] Munoz-Villegas P, Navarro-Sanchez AA, Sanchez-Rios A, Olvera-Montano O, Baiza-Duran LM. Reexamining Ophthalmic Drugs, Safety and Tolerability in Phase 1 Clinical Trials. Ther Clin Risk Manag. 2021 Oct 21;17:1123-1134. doi: 10.2147/TCRM.S331294. eCollection 2021. PMID 34707360

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Lagricel® Ofteno Multidose: Lagricel® Ofteno Multidose 0.4% hyaluronate. Ophthalmic solution. Laboratorios Sophia
  lagricel ofteno multidose: - Dosage: 1 drop 4 times a day per 7 days, both eyes
  - Route of administration: Ophthalmic
- Lagricel® Ofteno Single Dose: Lagricel® Ofteno single dose. 0.4% hyaluronate. Ophthalmic solution. Laboratorios Sophia
  lagricel ofteno single dose: - Dosage: 1 drop 4 times a day per 7 days, both eyes
  - Route of administration: Ophthalmic
Period: Overall Study
Arm/Group | Lagricel® Ofteno Multidose | Lagricel® Ofteno Single Dose
Started | 16; 32 Eyes | 18; 36 Eyes
Completed | 16; 32 Eyes | 18; 36 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lagricel® Ofteno Multidose | Lagricel® Ofteno Single Dose | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (6.6) | 29.7 (7.9) | 29.0 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 4 | 9 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Presence of Adverse Events (AEs)
Description: the adverse events will be evaluated with a scale of Present / Absent, it is a nominal variable, the normal value is absent
Time Frame: during the 10 days of evaluation, including the safety call (day 11).
Measure: Count of Participants; unit: Participants
Arm/Group | Lagricel® Ofteno Multidose | Lagricel® Ofteno Single Dose
Number analyzed (Participants) | 16 | 18
Participants | 7 | 8
Statistical Analysis 1: Comparison: Lagricel® Ofteno Multidose vs Lagricel® Ofteno Single Dose; Test type: Non-Inferiority — Compare the safety of the Lagricel® Ofteno multi-dose formulation against Lagricel® Ofteno unit doses manufactured by Sophia Laboratories S.A. of C.V. through the incidence of AD; p = 0.409, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.05

2. Primary Outcome: Eye Comfort Index (ECI)
Description: It is a questionnaire designed to measure the irritation of the ocular surface with Rasch analysis to produce estimates on a linear scale of intervals (ratings: 0-100).The Eye comfort index contains items that focus on the discomfort associated with alterations of the ocular surface.(0: None discomfort, 100: high discomfort).
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lagricel® Ofteno Multidose | Lagricel® Ofteno Single Dose
Number analyzed (Participants) | 16 | 18
score on a scale
  Inicial ECI | 29.98 [20.31 to 39.66] | 27.28 [21.38 to 33.18]
  Final ECI | 18.76 [12.31 to 25.21] | 18.01 [11.57 to 24.44]
Statistical Analysis 1: Comparison: Lagricel® Ofteno Multidose vs Lagricel® Ofteno Single Dose; Test type: Non-Inferiority — Compare the tolerability of the Lagricel® Ofteno multi-dose formulation against Lagricel® Ofteno unit-dose manufactured by Sophia Laboratories S.A. of C.V. using the ICO score; p = 0.442, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Lagricel® Ofteno Multidose; Final vs initial Eye Comfort Index; Test type: Equivalence — F=2.606, 15.926; p = 0.009, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Lagricel® Ofteno Single Dose; Final vs initial Eye Comfort Index; Test type: Equivalence — F=3.051, 19.336; p = 0.002, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Visual Acuity (VA)
Description: Visual acuity (VA) is a test of visual function. It will be evaluated at baseline, without refractive correction with the Snellen chart.Which will be located in a place with adequate lighting, natural or artificial and at a distance of 3meters from the subject to be evaluated. The snellen chart consists of a booklet with 11 lines composed of letters, each line has a different size and a different weighting. the subject is placed at a safe distance and the contralateral eye to which it will be evaluated is covered, then the examiner detects until the line can clearly see the letters given he or she a score, the normal score for a VA is 20/20.
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Lagricel® Ofteno Multidose | Lagricel® Ofteno Single Dose
Number analyzed (Participants) | 16 | 18
LogMAR
  Final VA | 0.988 (0.05) | 0.989 (0.05)
  Initial VA | 0.969 (0.09) | 0.989 (0.05)
Statistical Analysis 1: Comparison: Lagricel® Ofteno Multidose vs Lagricel® Ofteno Single Dose; Test type: Non-Inferiority — Compare the safety of the Lagricel® Ofteno multi-dose formulation against Lagricel® Ofteno unit doses manufactured by Sophia Laboratories S.A. of C.V. through changes in BCVA; p = 0.904, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Lagricel® Ofteno Multidose; Final vs initial VA; Test type: Equivalence — F=-1.414, 1.061; p = 0.157, Sign test
Statistical Analysis 3: Comparison: Lagricel® Ofteno Single Dose; Final vs initial VA; Test type: Equivalence; p = 1.000, Sign test

4. Secondary Outcome: Epithelial Defects (ED) Fluorescein Stain
Description: The epithelial defects will be evaluated by means of two stains, green lysine and fluorescein, it is a discrete variable that will be realized by direct observation, it will be staged according to the degrees of the oxford scale that go from 0 to 5 (0-V) according to its severity, where 0 is the normal lower limit and 5 the upper limit of defects.
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Population: Initial Fluorescein Staining Grade 0 (Lagricel® Ofteno Multidose n=22; Lagricel® Ofteno Single dose n=26) Initial Fluorescein Staining Grade 1 (Lagricel® Ofteno Multidose n=8; Lagricel® Ofteno Single dose n=8) Initial Fluorescein Staining Grade 2 (Lagricel® Ofteno Multidose n=2; Lagricel® Ofteno Single dose n=2)
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Lagricel® Ofteno Multidose | Lagricel® Ofteno Single Dose
Number analyzed (Participants) | 16 | 18
Number analyzed (Eyes) | 32 | 36
Eyes
  Final Fluorescein Staining Grade 0 | 30 | 34
  Final Fluorescein Staining Grade 1 | 2 | 2
Statistical Analysis 1: Comparison: Lagricel® Ofteno Multidose vs Lagricel® Ofteno Single Dose; Test type: Non-Inferiority — Compare the safety of the Lagricel® Ofteno multi-dose formulation against Lagricel® Ofteno unit doses manufactured by Sophia Laboratories S.A. of C.V. by changes in corneal and conjunctival staining with fluorescein; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Lagricel® Ofteno Multidose; Final vs initial fluorescein staining; Test type: Equivalence — Chi-squared (2)= 6.400; p = 0.041, Chi-squared
Statistical Analysis 3: Comparison: Lagricel® Ofteno Single Dose; Test type: Equivalence — Chi-squared (2)=0.814; p = 0.665, Chi-squared

5. Secondary Outcome: Epithelial Defects (ED) Green Lissamine
Description: as for outcome 4
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Population: Initial Lissamine Green Staining Grade 0 (Lagricel® Ofteno Multidose n=24; Lagricel® Ofteno Single dose n= 23 Initial Lissamine Green Staining Grade 1 (Lagricel® Ofteno Multidose n=6; Lagricel® Ofteno Single dose n= 11 Initial Lissamine Green Staining Grade 2 (Lagricel® Ofteno Multidose n=1; Lagricel® Ofteno Single dose n= 2 Initial Lissamine Green Staining Grade 3 (Lagricel® Ofteno Multidose n=1; Lagricel® Ofteno Single dose n= 0)
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Lagricel® Ofteno Multidose | Lagricel® Ofteno Single Dose
Number analyzed (Participants) | 16 | 18
Number analyzed (Eyes) | 32 | 36
Eyes
  Final Lissamine Green Staining Grade 0 | 29 | 31
  Final Lissamine Green Staining Grade 1 | 3 | 5
Statistical Analysis 1: Comparison: Lagricel® Ofteno Multidose vs Lagricel® Ofteno Single Dose; Test type: Non-Inferiority — Compare the safety of the Lagricel® Ofteno multi-dose formulation against Lagricel® Ofteno unit doses manufactured by Sophia Laboratories S.A. of C.V. by changes of corneal and conjunctival staining with lysamine green; p = 0.713, Fisher Exact
Statistical Analysis 2: Comparison: Lagricel® Ofteno Multidose; Final vs initial lissamine green staining; Test type: Equivalence — Chi-squared (3)=14.345; p = 0.002, Chi-squared
Statistical Analysis 3: Comparison: Lagricel® Ofteno Single Dose; Final vs initial lissamine green staining; Test type: Equivalence — Chi-squared (2)=0.506; p = 0.777, Chi-squared

6. Secondary Outcome: Conjunctival Hyperemia (CH)
Description: Conjunctival hyperemia will be evaluated as an ordinal variable, by direct observation and staged using the Efron scale as 0.-Normal / 1.-Very Light/ 2.- Light/ 3.-Mild / 4.-Moderate / 5.- Severe. Based on this scale, the normal and mild stages are considered without pathologies or normal. Mild, moderate and severe are considered pathological.
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Population: Initial conjunctival hyperemia (Lagricel® Ofteno Multidose n=26; Lagricel® Ofteno Single dose n=28)
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Lagricel® Ofteno Multidose | Lagricel® Ofteno Single Dose
Number analyzed (Participants) | 16 | 18
Number analyzed (Eyes) | 32 | 36
Eyes
  Hyperemia grade 0 (Normal) | 32 | 36
  Hyperemia grade 1 (Very Light) | 0 | 0
  Hyperemia grade 2 (Light) | 0 | 0
  Hyperemia grade 3 (Mild) | 0 | 0
  Hyperemia grade 4 (Moderate) | 0 | 0
  Hyperemia grade 5 (Severe) | 0 | 0
Statistical Analysis 1: Comparison: Lagricel® Ofteno Multidose vs Lagricel® Ofteno Single Dose; Test type: Non-Inferiority — Compare the safety of the Lagricel® Ofteno multi-dose formulation against Lagricel® Ofteno unit doses manufactured by Sophia Laboratories S.A. of C.V. by changes in conjunctival hyperemia; p = 1.000, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Lagricel® Ofteno Multidose; Final vs initial conjunctival hyperemia; Test type: Equivalence — F=4.167, 1; p = 0.031, Fisher Exact
Statistical Analysis 3: Comparison: Lagricel® Ofteno Single Dose; Final vs initial conjunctival hyperemia; Test type: Equivalence — No significant change was observed; p = 1.000, Chi-squared, Corrected

7. Secondary Outcome: Chemosis
Description: It is defined as conjunctival edema, the result of an inflammatory reaction. It is qualified as present or absent. The evaluator will use a narrow beam of light at 60 ° and will measure if the conjunctiva separates from the sclera by ≥ 1/3 of the total eyelid opening
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Population: Initial Chemosis (Lagricel® Ofteno Multidose, n=0; Lagricel® Ofteno Single dose, n=0)
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Lagricel® Ofteno Multidose | Lagricel® Ofteno Single Dose
Number analyzed (Participants) | 16 | 18
Number analyzed (Eyes) | 32 | 36
Eyes
  Final chemosis present | 0 | 0
  Final chemosis absent | 32 | 36

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the study, which lasted about 1 month and 15 days.
Arm/Group | Lagricel® Ofteno Multidose | Lagricel® Ofteno Single Dose
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 7/16 | 8/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lagricel® Ofteno Multidose (N=16) | Lagricel® Ofteno Single Dose (N=18)
blurred vision (Eye disorders) | 2 (2) | 3 (3)
burning eyes (Eye disorders) | 4 (4) | 5 (5)
eye itching (Eye disorders) | 2 (2) | 1 (1)
dysgeusia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Tearing (Eye disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
foreign body sensation (Eye disorders) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Only the sponsor has the decision to disseminate or publish the information obtained from the investigation and the PIs involved must submit a formal request to the sponsor if they are willing to disseminate or publish such information, they may only publish them if they have the written authorization of the sponsor (Laboratoios Sophia S.A. de C.V.).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT04081610/Prot_SAP_000.pdf